CLINICAL TRIAL: NCT06310967
Title: A Dose Escalation Study of IG3018 to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics in Subjects With Hyperuricemia With or Without Chronic Kidney Disease
Brief Title: A Dose Escalation Study of IG3018 in Subjects With Hyperuricemia With or Without Chronic Kidney Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intelligem Therapeutics Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IG3018-23-02-01
Record Dates: First submitted 2024-03-03; First posted 2024-03-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Hyperuricemia; Hypouricemia, Renal
Keywords: Hyperuricemia, Renal; Hyperuricemia; Chronic Kidney Disease; CKD; Hyperuricemia, CKD
MeSH Terms: conditions — Hyperuricemia; Renal hypouricemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Part 1 is a randomized, double-blind, placebo-controlled study where the doses of the study drug are escalated in a predesigned manner in 3 cohorts.
  Initiation Dose shall be at 0.25 g tablets (Cohort A) and doses are escalated to 0.5 g (Cohort B) and then to 1.0 g (Cohort C) in a planned manner. Each cohort will have 10 eligible patients. Randomization will be performed in Part 1 and as per the randomization code, 8 subjects will receive the active study drug (IG3018) and 2 shall receive placebo in each dose cohort. A total of 30 subjects are planned to be enrolled.
  Part 2 is an open-label PoC study involving hyperuricemia subjects with advanced predialysis CKD (Stage 3a, Stage 3b and Stage 4), and treated with two doses of IG3018 [0.5 g BID (Cohort D) and 1.0 g BID (Cohort E)]. 12 to 15 hyperuricemia subjects with advanced predialysis CKD (at least 6 Taiwanese subjects are required) will be enrolled in each dose and will receive the determined study dose of IG3018 BID for 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 is a randomized, double-blind, placebo-controlled study. For each dose cohort in Part 1, the Sponsor, subjects and other personnel involved with the conduct of the study will be blinded to the study products.
  Part 2 is an open-label proof of concept study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort A (0.25 g tablets) (Other): Cohort A will have 10 eligible patients. 8 subjects will receive the active study drug (IG3018) and 2 shall receive placebo in each dose cohort.
  Dose shall be at 0.25 g tablets. Single-dose initial treatment phase: D1~D3. Subject will receive a single dose of IG3018 or the placebo on Day 1. The predetermined information shall be collected in the form of blood and urine samples for PK analyses, whilst efficacy and safety assessment data will be collected within 48 hours after the single dose of study drug administration (IG3018 or placebo).
  Maintenance treatment on daily basis phase: 4 weeks. Subjects in this maintenance treatment phase shall receive the study drug IG3018 in twice daily dosing for 28 days from Day 4 to Day 31, and will be given IG3018 once on the morning of D32.
  Interventions: Drug: IG3018; Other: Placebo matching IG3018
- Cohort B (0.5 g tablets) (Other): Cohort B will have 10 eligible patients. 8 subjects will receive the active study drug (IG3018) and 2 shall receive placebo in each dose cohort.
  Dose shall be at 0.5 g tablets. Single-dose initial treatment phase: D1~D3. Subject will receive a single dose of IG3018 or the placebo on Day 1. The predetermined information shall be collected in the form of blood and urine samples for PK analyses, whilst efficacy and safety assessment data will be collected within 48 hours after the single dose of study drug administration (IG3018 or placebo).
  Maintenance treatment on daily basis phase: 4 weeks. Subjects in this maintenance treatment phase shall receive the study drug IG3018 in twice daily dosing for 28 days from Day 4 to Day 31, and will be given IG3018 once on the morning of D32.
  Interventions: Drug: IG3018; Other: Placebo matching IG3018
- Cohort C (1.0 g tablets) (Other): Cohort C will have 10 eligible patients. 8 subjects will receive the active study drug (IG3018) and 2 shall receive placebo in each dose cohort.
  Dose shall be at 1.0 g tablets. Single-dose initial treatment phase: D1~D3. Subject will receive a single dose of IG3018 or the placebo on Day 1. The predetermined information shall be collected in the form of blood and urine samples for PK analyses, whilst efficacy and safety assessment data will be collected within 48 hours after the single dose of study drug administration (IG3018 or placebo).
  Maintenance treatment on daily basis phase: 4 weeks. Subjects in this maintenance treatment phase shall receive the study drug IG3018 in twice daily dosing for 28 days from Day 4 to Day 31, and will be given IG3018 once on the morning of D32.
  Interventions: Drug: IG3018; Other: Placebo matching IG3018
- Cohort D (0.5 g BID IG3018) (Other): 12 to 15 hyperuricemia subjects with advanced predialysis CKD (at least 6 Taiwanese subjects are required) will be enrolled in Cohort D and will receive 0.5 g IG3018 twice daily (BID) for 4 weeks.
  Interventions: Drug: IG3018
- Cohort E (1.0 g BID IG3018) (Other): 12 to 15 hyperuricemia subjects with advanced predialysis CKD (at least 6 Taiwanese subjects are required) will be enrolled in Cohort E and will receive 1.0 g IG3018 twice daily (BID) for 4 weeks.
  Interventions: Drug: IG3018

INTERVENTIONS:
Drug: IG3018 — Oral administration
Other: Placebo matching IG3018 — Oral administration
  Arms: Cohort A (0.25 g tablets); Cohort B (0.5 g tablets); Cohort C (1.0 g tablets)

SUMMARY:
This is a phase I/II clinical study to evaluate the safety, tolerability, PK, and efficacy of IG3018 tablet in hyperuricemia (HUA) subjects with or without CKD.

DETAILED DESCRIPTION:
The study has two parts:

Part 1 is a randomized, double-blind, placebo-controlled, dose escalation study in hyperuricemia subjects without CKD. Initiation Dose shall be at 0.25 g tablets (Cohort A) and doses are escalated to 0.5 g (Cohort B) and then to 1.0 g (Cohort C) in a planned manner.

Part 2 is an open-label, proof of concept study involving hyperuricemia subjects with advanced predialysis CKD (Stage 3a, Stage 3b and Stage 4), and treated with two doses [0.5 g BID IG3018 (Cohort D) and 1.0 g BID IG3018 (Cohort E)].

ELIGIBILITY:
Inclusion Criteria:

For Part 1 and Part 2:

Subjects must meet all the following criteria to be included in the study:

1. Male or female, aged 18 to 75 years (both inclusive).
2. According to the investigator's judgment, eGFR must be met as:

   Part 1 only: subjects without CKD and have eGFR ≥ 60 mL/minute/1.73 m2 at screening phase; Part 2 only: subjects with advanced predialysis CKD (Stage 3a, 3b and Stage 4) have eGFR≥15 and <60 mL/minute/1.73 m2 at screening phase.
3. The serum uric acid level for subjects need to meet any of the following:

   For subjects already on ULT within 2 weeks prior to the screening visit, the serum uric acid would be measured during the screening visit/phase, and then at the end of the run-in phase, prior to confirming their eligibility. Subjects with ULT within 2 weeks before screening has fasting serum uric acid ≥ 0.48 mmol/L at the end of run-in phase.

   For subjects without ULT in 2 weeks prior to screening visit，the serum uric acid should be measured twice on 2 different days (at least 24 hours apart) prior to confirming their eligibility. Subjects without ULT within 2 weeks before screening has fasting serum uric acid ≥ 0.48 mmol/L at screening phase.
4. Body Mass Index (BMI) ≥ 18 and ≤ 35 kg/m2 (both inclusive) at screening.
5. Female subjects of child-bearing potential [defined as women who have experienced menarche but have not reached postmenopausal status (defined as at least 12 consecutive months of amenorrhea without any other identifiable cause other than menopause), and who have not undergone surgery (i.e., bilateral oophorectomy and/or bilateral salpingectomy and/or hysterectomy) or have no other cause of permanent infertility as determined by the investigator (e.g., Müllerian agenesis).] must agree to use highly effective contraceptive methods and must abstain from egg collection or donation from the screening phase to 90 days after the last dose of the IMP. And the male partner of a female subject also needs to agree to use highly effective method of birth control during this phase.
6. Male subjects considered fertile must agree to not donate sperm, and take effective contraceptive methods from the screening phase to 90 days after the last dose of the IMP. And the female partner of male subjects also needs to agree to use a highly effective method of female contraception during this phase.
7. Able to understand and give signed written informed consent form (ICF) and willing to comply with all study procedures.

   Only for Part 2
8. For subjects with anemia who require iron supplementation, steady iron or iron-containing drugs should be used for at least 3 months, and the original treatment regimen should be maintained during the study period.

Exclusion Criteria:

For Part 1 and Part 2:

Subjects who meet any of the following criteria will be excluded from the study:

1. Prior uricase/recombinant uricase (such as Rasburicase or Pegloticase) therapy within 2 weeks prior to screening or last dose of therapy< 5 times the half-life (whichever is longer).
2. Subjects who have acute gout flares requiring treatment within 4 weeks prior to or during screening.
3. Major surgery within 3 months prior to the first administration.
4. History of malignant tumors within 6 months prior to screening.
5. Subjects within the last 3 months have: myocardial infarction, angina, percutaneous transluminal coronary angioplasty, coronary artery bypass grafting, cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, or transient ischemia attack.
6. Subjects who are on other urate-lowering medication (allopurinol, febuxostat, probenecid and benzbromarone) and cannot stop during the study periods included in the run-in phase.
7. Subject with underlying medical conditions requiring changes or introduction of drugs that have the potential impact on the serum uric acid levels (e.g., salicylic acids, diuretics, angiotensin receptor blockers, etc.) within at least 1 month prior the screening phase.
8. History of gastrointestinal (GI) surgery, including gastric sleeve, colostomy/enterostomy, Roux-en-Y or gastric banding (unless gastric band removed for a minimum of 12 months prior to screening.
9. History of GI diseases, including gastrointestinal bleeding moderate to severe gastrointestinal dysfunction, moderate to severe chronic constipation for a minimum of 3 months prior to screening, or newly diagnosed peptic or duodenal ulcer diseases within 4 weeks prior to screening.
10. Chronic use of parenteral nutrition including manganese within 3 months prior to screening.
11. Subjects who have the history of manganese toxicity or excessive exposure to manganese (i.e., having worked in a mine, foundry, smelter, dry cell battery manufacturing facility) within 2 months prior to screening.
12. Inability to swallow oral medications.
13. Received treatment with or exposure to an investigational drug or device within 30 days of signing informed consent.
14. Subjects with one of positive results of HIV virus or syphilis, or positive hepatitis B virus surface antigen (HBsAg) and the number of copies of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) ≥ 500 IU/mL (or 2500 copies, or the lower limit of the positive detection value of the study site) at screening, or HBsAg (-), hepatitis B core antibody (HBcAb) (+) and the number of copies of HBV DNA ≥ 500 IU/mL (or 2500 copies, or the lower limit of the positive detection value of the study site) after treatment of HBV infection, or positive hepatitis C antibody (HCV-Ab), and hepatitis C virus (HCV) ribonucleic acid (RNA) ≥upper limit of normal (ULN) of the study site during screening phase.
15. History of alcohol abuse, or subjects who consumed alcohol within 48 h before the first administration or did not agree to stop using alcohol products during the study.
16. Subjects who have previously been diagnosed with the following diseases and have not been able to control them after medication therapy or other treatment. Uncontrolled is defined as hypertension: sSBP ≥ 180 mmHg and/or sDBP ≥ 110 mmHg; or Diabetes mellitus: HbA1c ≥ 9% at screening.
17. Subjects with secondary hyperuricemia caused by tumor, hematological system diseases, drugs, etc. except for chronic kidney disease; or hereditary hyperuricemia at screening.
18. Subjects undergone kidney transplantation or planning to undergo kidney transplantation at screening.
19. Subjects with abnormal biliary function, biliary obstruction, or biliary gallstone at screening; Subjects with alanine aminotransferase (ALT) ≥3 ULN, aspartate aminotransferase (AST)≥3 ULN, or total bilirubin (TBIL) ≥1.5 ULN at screening.
20. Prior or current cholestatic liver disease defined as a clinical condition associated with decrease in bile flow due to impaired secretion by hepatocytes or to obstruction of bile flow through intra-or extrahepatic bile ducts.
21. History of serious hypersensitivity reaction to a known ingredient of IG3018 tablet judged by the investigator.
22. Subjects who are considered unsuitable for participating in the study in the opinion of the investigator judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Safety Assessments (Part 1 and Part 2) | Baseline through study completion at up to 46 days
  Safety as assessed by incidence of reported adverse events, clinically significant changes in vital signs, physical examination, laboratory tests, 12-lead ECG.
  Safety as assessed by incidence of AEs by using the Common Terminology Criteria for Adverse Events, Version 5 (CTCAEv5).
The proportions of change from baseline in serum uric acid to normal level (≤ 0.36 mmol/L) (Part 1 and Part 2) | 4 weeks
  The proportions of change from baseline in serum uric acid to normal level (≤ 0.36 mmol/L) following 4 weeks treatment with IG3018 in each dose.

SECONDARY OUTCOMES:
The proportions of change from baseline in serum uric acid to ≤ 0.30 mmol/L and ≤ 0.24 mmol/L respectively (Part 1 and Part 2) | 4 weeks
  The proportions of change from baseline in serum uric acid to ≤ 0.30 mmol/L and ≤ 0.24 mmol/L respectively, following 4 weeks treatment with IG3018 in each dose.
The actual change of serum uric acid (Part 1 and Part 2) | 4 weeks
  The actual change of serum uric acid from baseline to the end of 1, 2, 3, and 4 weeks of each treatment group.
The percentage change of serum uric acid (Part 1 and Part 2) | 4 weeks
  The percentage change of serum uric acid from baseline to the end of 1, 2, 3, and 4 weeks of each treatment group.
Gouty Attacks (Part 1 and Part 2) | Baseline through study completion at up to 46 days
  Incidence of reported gouty attacks during the study period.
Urinary Albumin/Creatinine Ration (U-ACR) (Part 2 only) | Baseline through study completion at up to 43 days
  The change in Urinary Albumin/Creatinine ration (U-ACR) during the study period.
Ae of IG3018 (Part 1 only) | 32 days
  Urine Accumulative excretion (Ae) of IG3018
Cmax of IG3018 (Part 1 only) | 46 days
  Maximum observed whole blood concentration of IG3018
Tmax of IG3018 (Part 1 only) | 46 days
  Time to reach maximum whole blood concentration of IG3018
T1/2 of IG3018 (Part 1 only) | 46 days
  Terminal half-life of IG3018
Estimated glomerular filtration rate (eGFR) (Part 2 only) | Baseline through study completion at up to 43 days
  The change in estimated glomerular filtration rate (eGFR) during the study period.
Cmax of IG3018 (Part 2 Taiwanese subjects only) | 43 days
  Maximum observed whole blood concentration of IG3018
Tmax of IG3018 (Part 2 Taiwanese subjects only) | 43 days
  Time to reach maximum whole blood concentration of IG3018
T1/2 of IG3018 (Part 2 Taiwanese subjects only) | 43 days
  Terminal half-life of IG3018

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (3):
  - Emeritus Research Pty Ltd -Sydney, Botany, New South Wales
  - Pendlebury Research Pty Ltd T/A Novatrials, Kotara, New South Wales
  - Emeritus Research Pty Ltd -Melbourne, Camberwell, Victoria
- Taiwan (3):
  - Chung Shan Medical University Hospital, Taichung, Taiwan
  - Taipei Medical University Hospital, Taipei, Taiwan
  - Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided